CLINICAL TRIAL: NCT00667966
Title: Double-blind, Cross-over, Placebo Controlled Pilot Study to Characterize the Profile of Those Patients With Spinal Cord Injury Diagnosed by Electrophysiological, Urodynamic and Clinical (ASIA Group) Assessment Who May Respond to Vardenafil Treatment. (LEMDE)
Brief Title: Assess Efficacy in Subjects With Traumatic Spinal Cord Injury
Acronym: LEMDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11861; 2004-005282-37 (EudraCT Number)
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Erectile Dysfunction; Spinal Cord Injury
Keywords: Spinal cord injury; Urodynamic; Erectile dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction; Spinal Cord Injuries | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vardenafil + Placebo (Experimental): Subjects received single dose of 10 mg vardenafil followed by 20 mg vardenafil and then crossed over to 10 mg placebo followed by 20 mg placebo.
  Interventions: Drug: Vardenafil (Levitra, BAY 38-9456), 10 mg; Drug: Placebo; Drug: Vardenafil (Levitra, BAY 38-9456), 20 mg
- Placebo + Vardenafil (Experimental): Subjects received single dose of 10 mg placebo followed by 20 mg placebo and then crossed over to 10 mg vardenafil followed by 20 mg vardenafil.
  Interventions: Drug: Vardenafil (Levitra, BAY 38-9456), 10 mg; Drug: Placebo; Drug: Vardenafil (Levitra, BAY 38-9456), 20 mg

INTERVENTIONS:
Drug: Vardenafil (Levitra, BAY 38-9456), 10 mg — 10 mg vardenafil was administered with a glass of water 1 h before starting the test with the stimulator.
Drug: Placebo — 10/20 mg placebo in sequence in respective arm
Drug: Vardenafil (Levitra, BAY 38-9456), 20 mg — 20 mg vardenafil was administered with a glass of water 1 h before starting the test with the stimulator.

SUMMARY:
Assess efficacy of Vardenafil in patients with traumatic spinal cord injury

ELIGIBILITY:
Inclusion Criteria:

* Men between 18 and 64 years old with stable cord injury (more than 6 months) who had erectile dysfunction according to the National Institutes if Health (NIH) after their traumatic spinal cord injury

Exclusion Criteria:

* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life-threatening arrhythmia within prior 6 month
* Nitrate therapy

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2005-07; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Characteristics of responders and non responder with respect to the electrophysiological (skin sympathetic response, bulbocavernosus reflex and somatosensory and pudendal evoked potential), urodynamical and clinical (ASIA group) tests | 4 treatment days
  Responders are defined as subjects with rigidity ≥ 60% in the base measured with RigiScan during at least 5 minutes after withdrawing the vibrator and/or finishing manual stimulation.

SECONDARY OUTCOMES:
Duration of an erection ≥ 60% in the base induced by an erectogenic stimulus (vibrator and/or manual) in each subject after administering a 10 mg dose of vardenafil or placebo | 4 treatment days
Duration of an erection ≥ 60% in the base induced by an erectogenic stimulus (vibrator and/or manual) in each subject after administering a 20 mg dose of vardenafil or placebo | 4 treatment days
Number of participants with adverse events | Approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Spain (2):
  - Badalona, Barcelona
  - Toledo, Toledo

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/